CLINICAL TRIAL: NCT05108662
Title: Comparison of Surgical Stress in Patients Undergoing TURP Versus HOLEP Surgery by Measuring Perioperative Systemic Inflammatory Markers
Brief Title: Inflammatory Markers: HOLEP Versus TURP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adana City Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Baris Arslan, MD, Baris Arslan, MD, Principal investigator, Adana City Training and Research Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 49-708
Record Dates: First submitted 2021-09-22; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Prostate Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HOLEP (Active Comparator): Patients with a prostate volume greater than 80 g
  Interventions: Procedure: Surgery method
- TURP (Active Comparator): Patients with a prostate volume less than 80 g
  Interventions: Procedure: Surgery method

INTERVENTIONS:
Procedure: Surgery method — Patients were subdivided into two groups according to their prostate volume

SUMMARY:
Aim of the study is to compare the systemic inflammatory markers and surgical stress response in patients undergoing HOLEP or TUR-P surgery.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) is the most common disease in aging men worldwide, causing significant difficulties and resulting in bladder outlet obstruction. Basically, surgical techniques in patients with BPH are transurethral resection of the prostate (TURP), holmium laser enucleation of the prostate (HOLEP), and open prostoactemy surgery. There are many studies comparing the clinical outcomes of TURP and HOLEP surgery. However, to the best of our knowledge, there has not been a study comparing the effects of these two types of surgery on inflammatory markers and stress hormones.

ELIGIBILITY:
Inclusion Criteria:

* ASA scores I-III patients
* having benign prostatic hyperplasia
* undergoing HOLEP or TURP surgery under general anesthesia

Exclusion Criteria:

* immune system disease,
* diabetes mellitus,
* malignancy other than prostate disease,
* history of steroid use,

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
inflamatory markers | Change from baseline WBC (109 /L) at postoperative 0th and postoperative 24th hour
  WBC (109 /L)
Stress hormone levels | Change from baseline adrenaline (ng/L) at postoperative 0th and postoperative 24th hour
  Adrenaline (ng/L)
inflamatory markers | Change from baseline CRP (mg/L) at postoperative 0th and postoperative 24th hour
  CRP
inflamatory markers | Change from baseline IL-6 (pg/ml) and TNF-alfa (pg/ml), at postoperative 0th and postoperative 24th hour
  IL-6 (pg/ml) and TNF-alfa (pg/ml)
inflamatory markers | Change from baseline CD4+/CD8+ at postoperative 0th and postoperative 24th hourL-6 (pg/ml) and TNF-alfa (pg/ml)
  CD4+/CD8+
stress hormone levels | Change from baseline cortisol (microg/dl) at postoperative 0th and postoperative 24th hour
  Cortisol (microg/dl)

CONTACTS AND LOCATIONS:
Overall Officials: Baris Arslan, MD, Principal Investigator — Adana City Training and Research Hospital
Locations (1):
- Adana City Training and Research Hospital, Adana, Turkey (Türkiye)